# STATISTICAL ANALYSIS PLAN

For:

Grifols Therapeutics LLC.

#### SPONSOR PROTOCOL No. GC1703

A Prospective, Open-Label, Single-Arm Clinical Trial to Assess the Anti-Hepatitis A Virus (HAV) Antibody Levels, Pharmacokinetics, and Safety of a Single Intramuscular Dose of a Polyvalent Human Immune Globulin in HAV-Seronegative Healthy Subjects





Version: FINAL 1.0

Date: 2018/04/24



We have carefully read this Statistical Analysis Plan and agree it contains the necessary information required to handle the statistical analysis of study data.



On behalf of the Sponsor:



# **VERSION CONTROL**

| Version<br>Number | Version Date | Author | Description of Significant Changes from Previous Approved Version |
|---|---|---|---|
| DRAFT 0.1 | 2018/02/12 | | Not Applicable – First Version |
| DRAFT 0.2 | 2018/03/16 | | Second version after first round of comments. Mock shells were added |
| DRAFT 0.3 | 2018/04/06 | | Third version after second round of comments |
| DRAFT 0.4 | 2018/04/19 | | Fourth version after third round of comments |
| FINAL 1.0 | 2018/04/24 | | Final Version |

# **CONTENTS**

| STATISTICAL ANALYSIS PLAN APPROVAL | | 2 |
|---|---|---|
| VERSION CONTROL | | 3 |
| ABBREVIATIONS | | 6 |
| 1. INTRODUCTION | | 8 |
| 2. STUDY OBJECTIVES Primary Efficacy Objective Pharmacokinetic (PK) Objectives Safety Objective | 9<br>9<br>9 | 9 |
| 3. STUDY DESIGN General Description Treatment Study procedures Randomization and Unblinding Procedures | 10<br>10<br>10<br>11 | 10 |
| 4. STUDY ENDPOINTS Efficacy Endpoints Pharmacokinetic Endpoints Safety Endpoints Sample Size Determination | 12<br>12<br>12<br>12 | 12 |
| 5. ANALYSIS POPULATIONS Safety Population Evaluable Population Pharmacokinetic Population | 13<br>13<br>13 | 13 |
| 6. STATISTICAL METHODOLOGY Analysis Timepoints Methods for Handling Missing Data | 14<br>14 | 14 |
| 7. STUDY SUBJECTS Disposition Protocol Deviations | 15<br>15 | 15 |
| 8. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS Demographic and Baseline Characteristics Medical History Contraceptive Methods Electrocardiogram | 16<br>16<br>16<br>16 | 16 |
| 9. EFFICACY Analysis of Anti-HAV Antibody Endpoint(s) | 17 | 17 |
| 10. PHARMACOKINETICS Analysis of Pharmacokinetic Endpoint(s) | 18 | 18 |
| 11. SAFETY Adverse Events Prior and Concomitant Medications Extent of Exposure Clinical Laboratory Evaluations | 21<br>21<br>22<br>22 | 21 |

| Vital Signs | 23 |
|-------------------------------------------------------|----|
| Physical Examination Findings | 24 |
| 12. INTERIM ANALYSES AND DATA SAFETY MONITORING | 25 |
| 13. CHANGES TO PROTOCOL-SPECIFIED ANALYSES | 26 |
| 14. GENERAL INFORMATION RELATED TO DATA PRESENTATIONS | 27 |
| PLANNED TABLES | 28 |
| PLANNED FIGURES | 29 |
| PLANNED LISTINGS | 29 |
| APPENDIX A | 3′ |
| STUDY SCHEDULES | 31 |
| APPENDIX B | 34 |
| TABLE SHELLS | 34 |
| APPENDIX C | 60 |
| LISTING SHELLS | 60 |
| APPENDIX D | 74 |
| SHELLS (FROM WINNONLIN) | 74 |

#### **ABBREVIATIONS**

ADR Adverse Drug Reaction

AE Adverse Event
Anti-HAV Anti-Hepatitis A Virus
ALP Alkaline Phosphatase
ALT Alanine Aminotransferase

aPTT Activated Partial Thromboplastin Time

AR Adverse Reaction

AST Aspartate Aminotransferase
ATC Anatomical/Therapeutic/Chemical

AUC<sub>0-∞</sub> Area under the serum concentration time curve extrapolated to infinity

AUC<sub>0-T</sub> Cumulative area under the or serum concentration time curve calculated from 0 to time of

last observed quantifiable serum concentration

BLQ Below Limit of Quantitation

BMI Body Mass Index
BUN Blood Urea Nitrogen
CI Confidence Interval

Cl<sub>TOT</sub>/F Apparent total serum clearance

C<sub>max</sub> Maximum observed serum concentration

CRF Case Report Form
CS Clinically Significant
CSR Clinical Study Report
CV Coefficient of Variation
DNA DeoxyriboNucleic Acid
ECG Electrocardiogram

GGT Gamma-glutamyl Transferase

HAV Hepatitis A Virus
HBV Hepatitis B virus
HCV Hepatitis C virus

HIV Human Immunodeficiency Virus

IM Intramuscular

IP Investigational Product

 $\lambda_z$  Apparent elimination rate constant

LDH Lactate Dehydrogenase

Max Maximum

MedDRA Medical Dictionary for Regulatory Activities

Min Minimum

NAT Nucleic Acid Test

NCA Non-compartmental Analysis

NCS Not Clinically Significant PΕ Physical Examination PΚ Pharmacokinetic(s) PΤ Prothrombin Time RNA RiboNucleic Acid SAE Serious Adverse Event SAP Statistical Analysis Plan SD Standard Deviation SOC System Organ Class

TEAE Treatment-Emergent Adverse Event

T<sub>half</sub> Terminal elimination half-life

 $T_{\text{max}}$  Time of maximum observed serum concentration

TFLs Tables, Figures, and Listings

WHO-DDE World Health Organization Drug Dictionary Enhanced

 $V_D/F$  Apparent volume of distribution

# 1. INTRODUCTION

This statistical analysis plan (SAP) provides a detailed description of the statistical methods and procedures to be implemented for the analyses of data to support the completion of the clinical study report (CSR). The analyses described in the SAP are based upon the final protocol GC1703/Protocol Version 5.0, dated 2018/01/22. Additional post-hoc or unplanned analyses, which are not defined in this SAP, may be performed to support the clinical development program. Such analyses will be documented in the CSR.

#### 2. STUDY OBJECTIVES

#### Primary Efficacy Objective

The primary efficacy objective is to evaluate whether a single 0.2 mL/kg intramuscular (IM) dose of the study treatment will provide protective levels of antibodies to Hepatitis A Virus (anti-HAV) in HAV-seronegative healthy subjects for up to 60 days.

#### Pharmacokinetic (PK) Objectives

The pharmacokinetic objectives are to evaluate the PK parameters of anti-HAV antibodies following a single 0.2 mL/kg IM dose of the study treatment in HAV-seronegative healthy subjects.

The PK parameters of interest are:

- Area under the serum concentration time curve extrapolated to infinity (AUC<sub>0-∞</sub>)
- Cumulative area under the serum concentration time curve calculated from 0 to time of last observed quantifiable serum concentration (AUC<sub>0-T</sub>)
- Maximum observed serum concentration (C<sub>max</sub>)
- Time of maximum observed serum concentration (T<sub>max</sub>)
- Apparent elimination rate constant  $(\lambda_z)$
- Terminal elimination half-life (Thalf)
- Apparent total serum clearance (Cl<sub>TOT</sub>/F)
- Apparent volume of distribution (V<sub>D</sub>/F)

#### Safety Objective

The safety objective is to evaluate the safety and tolerability of a single 0.2 mL/kg IM dose of the study treatment in HAV-seronegative healthy subjects.

#### 3. STUDY DESIGN

#### **General Description**

This is a single center, open-label, single-arm study. Approximately 28 HAV-seronegative healthy subjects will be enrolled and treated after obtaining their written informed consents. There will be a screening period of up to 28 days during which subjects will be screened for enrollment. Subjects will be male and 18 to 55 years of age, or female and 18 to 65 years of age, inclusive; and will weigh at least 50 kg at screening with a body mass index (BMI) of 18.5 to 29.9 kg/m². The healthy subjects will receive a single IM dose of GamaSTAN (0.2 mL/kg), which is followed by a PK sampling period of 150 days (approximately 5 half-lives). The protective levels of anti-HAV antibodies will be assessed up to 60 days after the administration of GamaSTAN. A PK curve will be obtained during the PK sampling period.

#### Treatment

A single 0.2 mL/kg IM dose of GamaSTAN [Immune Globuin (Human)] will be administered in the anterolateral aspects of the upper thigh or the deltoid muscle of the upper arm. Doses over 5 mL are to be divided and injected into several muscle sites to reduce local pain and discomfort.

#### Study procedures

The study consists of a Screening Visit, Treatment and Follow-up Visits, and Final Visit / Early Discontinuation Visit. Subjects will be qualified by screening assessments and procedures for reporting to the clinical site on Day -1. Subjects will be discharged from the clinic on Day 2, following the scheduled assessments and procedures, and will return to the clinical site for the remaining ambulatory PK samples and safety monitoring, and again for the final visit (Day 150). The total duration of study participation for subjects who complete the study will be approximately 178 days. For complete details on the study procedures and events, refer to Appendix A. The overall study schema is presented below:



PK sampling visits will be conducted as close as possible to the exact time points. The PK sampling visits: Day 1: prior to study drug injection, 60 minutes (±10 minutes) post study drug injection and 12 hours post study drug injection (a window of ±1 hour is permitted); Day 2 (window of ±1 hour); Days 3, 4 and 5 (visits have a window of ±4 hours); Days 7, 10, and 14 (all 3 visits have a window of ±1 day); Days 21 and 28 (both visits have a window of ±2 days); Days 60, 79 and 115 (all 3 visits have a window of ±4 days); Day 150 (a window of ±7 days)



# Randomization and Unblinding Procedures

This is an open label, single arm study, so blinding is not applicable and subjects are not randomized.

#### 4. STUDY ENDPOINTS

#### **Efficacy Endpoints**

The primary efficacy endpoint is the proportion of subjects maintaining protective anti-HAV antibody levels (defined as anti-HAV antibody titer  $\geq$ 10 mIU/mL in serum) after  $T_{max}$  up to 60 days after study treatment administration.

#### Pharmacokinetic Endpoints

With respect to the PK endpoint, the parameters of interest for this study are:  $AUC_{0-\infty}$ ,  $AUC_{0-T}$ ,  $C_{max}$ ,  $T_{max}$ ,  $\lambda_z$ ,  $T_{half}$ ,  $CI_{TOT/F}$  and  $V_{D/F}$ .

#### Safety Endpoints

The safety endpoints will include a summary of the incidence of adverse events (AEs), serious adverse events (SAEs), suspected adverse drug reactions (ADRs) and adverse reactions (ARs), as well as descriptive summary and statistics of the safety parameters (clinical laboratory values, vital signs and physical examination findings).

### Sample Size Determination

Approximately 28 healthy subjects will be enrolled and treated in this study which will provide about 20 evaluable subjects based on approximately 30% dropout rate. The sample size is chosen based on clinical considerations but not on a formal sample size calculation.

# 5. ANALYSIS POPULATIONS

#### Safety Population

The safety population consists of all subjects who received any amount of investigational product (IP).

#### **Evaluable Population**

The evaluable population consists of all subjects who received the entire dose of IP and had no major protocol deviations that would impact the efficacy analysis up to Day 60. Any deviations from the protocol will be recorded and evaluated before database lock.

#### Pharmacokinetic Population

The PK population consists of all subjects who received the entire dose of the IP and who provided sufficient serum concentration data to facilitate calculation of PK parameters. Subjects who did not complete the PK sampling schedule may be included in the PK analysis only for the PK parameters that are judged not to be affected by the missing sample(s). This decision is to be documented and approved by the sponsor before the database lock.

#### 6. STATISTICAL METHODOLOGY

All analyses will be conducted using the SAS® software, version 9.4.Pharmacokinetic analyses will be performed using Phoenix WinNonlin version 6.3 or later.

Adverse events and medical history will be classified using standard Medical Dictionary for Regulatory Activities (MedDRA) terminology Version 20.1.

Prior and concomitant medications will be coded with the World Health Organization Drug Dictionary Enhanced (WHO-DDE) dictionary version March 1, 2017.

Unless otherwise specified, the data listings will include all dosed subjects up to the point of study completion or discontinuation; exceptions will be listings pertaining to a subset of subjects only (e.g., subjects with protocol deviations) or a subset of records/events (e.g., abnormal laboratory values).

Categorical variables will be summarized using the PROC FREQ procedure. Continuous variables will be summarized using the PROC UNIVARIATE procedure. For In-transformed endpoints, geometric mean, geometric standard deviation, and coefficient of variation will also be presented.

The following general comments also apply to all statistical analyses and data presentations:

- Duration variables will be calculated using the general formula: (end date start date) +1.
- If the reported value of a clinical laboratory parameter cannot be used in a statistical summary table (e.g., a character string is reported for a parameter of the numerical type), a coded value must be appropriately determined and used in the statistical analyses. In general, a value involving lower and upper limit of normal range such as '<10' or '≤5' will be treated as '10' or '5' respectively, and a value such as '>100' will be treated as '100'. However, the actual values as reported in the database will be presented in data listings.
- Individual subject listings of all data represented on the CRFs will be provided to facilitate the
  investigation of tabulated values and to allow for the clinical review of all efficacy, PK, and safety
  parameters.
- When non-PK assessments are repeated for a given time point, only the non-missing result which is the closest to the dosing time will be included in summary tables

The analyses described in this plan are considered a priori, in that they have been defined prior to database lock. Any analyses performed subsequent to database lock will be considered post hoc and exploratory. Post hoc analyses will be labeled as such in the corresponding statistical output and identified in the CSR.

#### **Analysis Timepoints**

Unless otherwise specified, the baseline value will be defined as the last non-missing evaluation prior to the administration of the IP.

#### Methods for Handling Missing Data

No imputations of values for missing data will be performed.

#### 7. STUDY SUBJECTS

Unless otherwise specified, summary tables for protocol deviations, demographics and other baseline characteristics will be presented for the Safety Population.

#### Disposition

Subject disposition will be summarized for all screened subjects who always include the re-screened subjects, including:

- Number of subjects screened (i.e., count of all unique subject numbers) and within that the number of subjects re-screened;
- Number of subjects not dosed: count of all qualifying unique subject numbers, including the initial failure of re-screened subjects who ended up being dosed or failures for both times;
- Number of subjects dosed;
- Number and percentage of dosed subjects who completed the study;
- Number and percentage of dosed subjects discontinued from the study by primary reason for discontinuation and overall;
- Number and percentage of dosed subjects included in each of the study populations

The percentages will be calculated using the number of subjects dosed as denominator.

A listing of all screened subject's disposition will be provided. A listing of subjects included in each of the analysis populations will also be provided.

#### **Protocol Deviations**

Protocol deviations will be identified during the study and evaluated before database lock. Protocol deviation criteria and severity will be summarized and listed.

#### 8. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

#### Demographic and Baseline Characteristics

Demographic data and baseline characteristics will be presented in a data listing and summarized in a table by analysis population. Subject demographics include sex, age, ethnicity, and race. Baseline characteristics include height, weight, and BMI.

Clinical lab assessments only performed at screening and/or baseline will be provided in data listings, including pregnancy test, urine alcohol and drug panel testing, IgA, virus safety testing, and coagulation.

#### Medical History

Any medical history findings will be recorded and presented in a listing.

#### Contraceptive Methods

Contraceptive methods will be presented in a subject listing.

#### Electrocardiogram

Electrocardiograms (ECGs) will occur at Screening and on Day -1 for eligibility evaluation before IP administration. All data will be listed. Values out of the normal range judged by an Investigator as clinically significant will be considered AEs.

# 9. EFFICACY

# Analysis of Anti-HAV Antibody Endpoint(s)

The percentage of subjects maintaining anti-HAV antibody levels  $\geq$ 10 mIU/mL after  $T_{max}$  up to Day 60 following study treatment administration will be summarized.

The efficacy analysis will be performed on the evaluable and safety populations.

#### 10. Pharmacokinetics

#### Analysis of Pharmacokinetic Endpoint(s)

PK analyses will be performed on the PK population.

#### **Concentration Data**

Below limit of quantitation concentrations (coded BLQ) will be treated as zero for descriptive statistics. In the case where concentrations for anti-HAV antibodies cannot be determined due to bioanalytical or clinical reasons, these values will be set to missing for the statistical and pharmacokinetic analysis and will not be included for subsequent analysis.

Pre-dose concentration will be used as baseline for calculation of baseline corrected levels of anti-HAV antibodies. Baseline correction will be performed by subtracting predose values from post-dose values.

The anti-HAV antibody levels during the PK sampling period (up to Day 150 following study treatment administration) will be listed

The individual serum concentration/time figures will be presented using the actual sampling times whereas the mean and median serum concentration/time figures will be presented using the nominal sampling times.

Descriptive statistics will be calculated at each individual scheduled time point. serum concentration data will be summarized using the following descriptive statistics: number of non-missing values (N), arithmetic mean, standard deviation (SD), 90% CI for mean, coefficient of variation (CV%), median, minimum (min), maximum (max), geometric mean. The actual elapsed time between IP administration and each PK blood sample draw will be calculated and presented in concentration listing. The PK parameter calculation for each subject will be based on the actual elapsed time instead of the scheduled time or nominal time.

The PK blood sampling schedule and nominal time are shown below:

| Study Day | Scheduled Time Points | Nominal Time (Hours) |
|-----------|---------------------------|----------------------|
| 1 | Prior to treatment | 0 |
| 1 | 60 minutes post treatment | 1 |
| 1 | 12 hours post treatment | 12 |
| 2 | 24 hours post treatment | 24 |
| 3 | 48 hours post treatment | 48 |
| 4 | 72 hours post treatment | 72 |
| 5 | 96 hours post treatment | 96 |
| 7 | Day 7 | 144 |
| 10 | Day 10 | 216 |
| 14 | Day 14 | 312 |
| 21 | Day 21 | 480 |
| 28 | Day 28 | 648 |
| 60 | Day 60 | 1416 |
| 79 | Day 79 | 1872 |

| 115 | Day 115 | 2736 |
|-----|---------|------|
| 150 | Day 150 | 3576 |

#### **Pharmacokinetic Parameters**

Below limit of quantitation concentrations (coded BLQ) will be treated as zero for noncompartmental analysis (NCA).

The PK parameters will be derived from the anti-HAV antibody baseline uncorrected and baseline corrected serum concentrations versus time using NCA, with Phoenix WinNonlin version 6.3 or later (Model 200–202 Extravascular). Parameters to be calculated are listed in the table below:

| C <sub>max</sub> | Maximum observed serum concentration |
|---|---|
| T <sub>max</sub> | Time of maximum observed serum concentration; if it occurs at more than one time point, $T_{\text{max}}$ is defined as the first time point with this value |
| TLQC | Time of last observed quantifiable serum concentration |
| AUC <sub>0-T</sub> | Cumulative area under the serum concentration time curve calculated from 0 to $T_{LQC}$ using the linear trapezoidal method, where $T_{LQC}$ represents time of last observed quantifiable serum concentration |
| AUC <sub>0-∞</sub> | Area under the serum concentration time curve extrapolated to infinity, calculated as AUC <sub>T</sub> + $C_{LQC}/\lambda_Z$ , where $C_{LQC}$ is the measured concentration at time $T_{LQC}$ |
| AUC%Extrap | Percentage of AUC <sub>0-∞</sub> due to extrapolation from T <sub>QLC</sub> to infinity |
| T <sub>LIN</sub> | Time point where the log-linear elimination phase begins |
| λz | Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration <i>versus</i> time curve |
| Thalf | Terminal elimination half-life, calculated as ln(2)/λz |
| V <sub>D</sub> /F | Apparent Volume of Distribution calculated as follows: $V_D / F = \left( \frac{Dose}{K_{el} * AUC_{\infty}} \right)$ Where Kel = $\lambda z$ . |
| СІтот/F | Apparent Total serum Clearance calculated as follows: $Cl_{TOT} / F = \left( \frac{Dose}{AUC_{\infty}} \right)$ |

Actual sampling times (hours, relative to the corresponding administration time) will be used for calculation of PK parameters. It is recognized that there may be circumstances where PK sampling may fall outside of the time windows.

In the case where less than 3 consecutive measurable concentrations of anti-HAV antibodies are observed, the AUC parameters will not be estimated for that specific profile for the analyte in question.

The main absorption and disposition parameters will be estimated using a non-compartmental approach with a log-linear terminal phase assumption. The linear trapezoidal rule will be used to estimate the area under the curve (linear trapezoidal linear interpolation) and the terminal phase will be estimated by maximizing the coefficient of determination estimated from the log-linear regression model. However,  $AUC_{0-\infty}$ ,  $\lambda_Z$ ,  $T_{half}$ ,  $CI_{TOT}/F$  and  $V_D/F$  parameters will be estimated for individual concentration-time profiles only when the terminal log-linear phase can be reliably characterized using the following criteria:

- Phoenix® WinNonlin® Best fit range selection (kel selection is to be reviewed and adjusted (time range) as appropriate)
- R<sup>2</sup> of at least 80%

Descriptive statistics for PK parameters of interest (AUC<sub>0...</sub>, AUC<sub>0.T</sub>, C<sub>max</sub>, T<sub>max</sub>,  $\lambda_z$ , T<sub>half</sub>, Cl<sub>TOT/F</sub> and V<sub>D/F</sub>) will be summarized using the following descriptive statistics: N, arithmetic mean, SD, 90% CI for mean, CV%, median, min, max, geometric mean (except T<sub>max</sub>), and 90% CI for geometric mean (except T<sub>max</sub>).

Additional PK parameters may be calculated if required.

#### **Data Precision**

Individual baseline uncorrected and baseline corrected PK concentrations will be displayed with the same precision used in the results from the bioanalytical laboratory.

Precision for individual PK parameters will be displayed with the same precision as per the bioanalytical results, except for the following:

- Observed PK parameters associated with time (e.g. T<sub>max</sub>, T<sub>LQC</sub>, T<sub>LIN</sub>) with 2 decimals places;
- Number of point (terminal phase characterization) with 0 decimal places;
- R<sup>2</sup> and λ<sub>z</sub> [Lambda z] with 4 decimal places;
- Percentages will be displayed with two decimal places.

Summary statistics for raw concentrations and PK parameters will be displayed with the same number of decimal places as the individual values unless specified otherwise

#### 11. SAFETY

Safety analyses will be performed on the safety population. Safety data will be summarized with descriptive statistics and frequency tables and will include clinical laboratory values, vital signs and physical examination findings. The incidence of AEs, suspected ADRs, ARs, and AEs by severity and causality will be summarized. Deaths, subjects with SAEs and AEs leading to premature discontinuation from the study will be listed and presented in narrative form.

#### **Adverse Events**

Suspected ADRs are the AEs with causality assessment of possibly or definitely related. Adverse reactions (ARs) are the AEs with causality assessment of definitely related.

Adverse events will be coded and classified using MedDRA® terms (system organ class and preferred terms). Adverse events will be classified as Treatment-Emergent Adverse Events (TEAEs) or non-TEAEs depending on the comparison of AE onset date/time with the start date/time of study treatment with the IP. A TEAE will be defined as an AE which occurs on or between the beginning of the study drug injection and the final visit of the clinical trial. A non-TEAE will be defined as an AE which occurs prior to the start of study treatment. For AEs with incomplete start dates, the same algorithm for missing or partial end date information described for prior and concomitant medication below will be used for determination of treatment emergent or not. Non-TEAEs and TEAEs will be summarized separately. All AEs will be summarized by presenting subject incidences and percentages, and they will also be listed by body systems with subject number. In addition, TEAEs, including suspected ADRs, will be summarized by system organ class, preferred term, causalrelationship, intensity (severity) and seriousness (serious vs non-serious) and injection site reactions (by severity and by location) using descriptive statistics. For the summary by severity or causality at each level of summarization (number of subjects, System Organ Class (SOC), or Preferred Term), a subject will only be counted once per system organ class or preferred term using the most severe AE or the AE with the strongest causal relationship to the IP. Subjects with an SAE or who withdraw from the study because of an AE will also be individually listed and summarized. In addition, a table summarizing the temporally-associated AEs defined as AEs happening during IP injection or within 24 hours following the end of IPinjection and within 72 hours following the end of IP injection will be presented.

In the overall summary table of TEAEs, the following will be presented:

- Number and percentage of subjects with TEAEs, total number of TEAEs;
- Number and percentage of subjects with suspected ADRs, total number of suspected ADRs;
- Number and percentage of subjects with ARs, total number of ARs;
- Number and percentage of subjects with SAEs, total number of SAEs;
- Number and percentage of subjects with AEs leading discontinuation from the study, total number of such events:
- Number and percentage of subjects with AEs with death as outcome, total number of such events;
- Number and percentage of subjects with injection site reactions, total number of such events
- Number and percentage of subjects with TEAEs during/within 24 Hours post end of IP injection
- Number and percentage of subjects with TEAEs during/within 72 Hours post end of IP injection

Subject listings of all AEs including severity and relationship to study drug, as well as the time from the injection start date will be provided. AEs leading to discontinuation from the study, SAEs, and deaths will also be presented in separate listings.

#### Prior and Concomitant Medications

Any prior and concomitant medications recorded will be presented in a data listing and summarized in a table.

Prior medications are those taken in the 30 days prior to screening visit and stopped before the start of the IP administration

Concomitant medications are defined as medications with a start date/time on or after the first study drug dosing, or ongoing or with an end date/time after the first dosing.

The following convention will be used for missing or partial end date information in order to determine whether a medication is prior or concomitant:

The unknown portions of a medication end date will be assumed to be as late as possible. If a medication end date is incomplete but the month/year of medication end date is prior to the month/year of the start of study treatment, then the medication will be considered a prior medication. If a medication end date is incomplete but the month/year of medication end date is the same as the month/year of the start of study treatment, then the medication will be considered a concomitant medication. All other incomplete medication end dates and all medications with missing end dates will be assumed to be concomitant medications.

The medication name, dose, units, route, formulation, frequency, indication or reason taken, any relationship to medical history or an AE, code, date and time taken will be presented. The start or end dates will be displayed in listings as recorded in CRF. The listing will include the coding terms (e.g., Anatomical/Therapeutic/Chemical terms (ATCs)).

The summary table will be sorted alphabetically by medication class (i.e., ATC Level 2) and medication sub-class (i.e., ATC level 4). If the ATC Level 4 term is missing, the ATC Level 3 term will be used in the medication summary table and data listing. For the summary tables, if a subject has taken a medication more than once, the subject will be counted only once at the ATC level.

#### **Extent of Exposure**

A listing summarizing date and time of study drug administration, dose administered, total volume prepared, route of administration, injection site, volume administered per site, needle size, total volume administered, percentage of volume administered (Volume Administered (mL)/ Volume Prepared (mL)\*100), and comments about dosing issues and deviations, where applicable, will be presented. A summary table of total volume prepared (mL), total volume administered (mL), treatment compliance (=total volume administered / total volume prepared x 100%), duration of treatment administration (minute), and injection site will be provided by analysis population as well.

#### **Clinical Laboratory Evaluations**

All clinical laboratory data (Table 1) will be listed for each subject. Complete results of each category of laboratory tests will be presented in respective listings. Clinical laboratory assessments will include hematology, chemistry, and urinalysis. Hematology panel: hemoglobin, hematocrit, platelets, red blood cell count, and white blood cell count (absolute and % with differential). Chemistry panel: Sodium, potassium, creatinine, blood urea nitrogen (BUN), calcium, lactate dehydrogenase (LDH), aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), glucose, total bilirubin, direct and indirect bilirubin. Urinalysis panel: Microscopic evaluation is done only with cause, pH, protein, glucose, and blood.

Subject listings of laboratory values will be provided. Values out of the normal range judged by an Investigator as clinically significant (CS) will be considered AEs. Summary tables of change from baseline and shift from baseline by visit will be provided for hematology, chemistry, and urinalysis. In addition, a summary of HAV ribonucleic acid (RNA) at baseline will be presented for all subjects.

Table 1: Name, Description, and Location of Laboratory Tests and Procedures

| Test Panel | Description | Location |
|---|---|---|
| Hematology | Hemoglobin, hematocrit, platelets, red blood cell count, white blood cell count (absolute and % with differential) | Central |
| Chemistry | Sodium, potassium, creatinine, calcium, BUN, LDH, AST, ALT, GGT, ALP, glucose, total bilirubin, direct and indirect bilirubin | Central |
| Coagulation <sup>1</sup> | Prothrombin time (PT) and activated partial thromboplastin time (aPTT) | Central |
| Immunoglobulin A (IgA) <sup>1</sup> | Quantitative | Central |
| Urine pregnancy test <sup>2</sup> | Qualitative urine β-HCG for female subjects | Local |
| Urine test for alcohol and drugs of abuse | Alcohol, marijuana, opiates, cocaine, amphetamines, methamphetamines, and benzodiazepines | Central |
| Urinalysis | Microscopic evaluation is done only with cause. | Central |
| | pH, protein, glucose and blood | |
| Virus safety (nucleic acid test | Screening: | |
| (NAT)) testing | HAV ribonucleic acid (RNA), Hepatitis B virus (HBV) DeoxyriboNucleic Acid (DNA), Hepatitis C virus (HCV) RNA, Human Immunodeficiency Virus (HIV)-1 RNA, and B19V DNA testing | Central |
| Virus safety (serology) testing | Screening: | |
| | hepatitis A antibody differential (IgM/IgG), hepatitis B core antibody differential (IgM/IgG), hepatitis C antibody, HIV-1/-2 + Group O antibody, and B19V antibody differential (IgM/IgG) testing | Central |
| Virus safety (NAT and serology) retain samples <sup>3</sup> | Day 1 prior to study drug injection and final visit | |

- 1. Screening visit only.
- 2. Screening and on Day -1, prior to study treatment administration.
- 3. Virus safety (NAT and serology) retain samples collected during the study will only be tested if subject exhibits clinical signs and symptoms consistent with HAV, HBV, HCV, HIV or B19V infection while participating in the study. Virus safety retain samples will be retained until all analyses in support of the study are complete.

#### Vital Signs

Blood pressure (systolic and diastolic), heart rate, respiratory rate and body temperature, will be measured at screening and on study Days -1, 1, 5, 28 and 60, and at final visit on Day 150 (or early discontinuation visit). Results of vital signs will be presented in a listing. Values out of the normal range judged by an Investigator as CS will be considered AEs. Summary table for change from baseline by visit will be provided.

# Physical Examination Findings

Physical examination (PE) includes a review of the following: head and neck, heart, lungs, abdomen and general appearance. This will occur at Screening visit and at final visit on Day 150 (or early discontinuation visit) for the complete PE, study Days -1, 2, 5, 28 and 60 for the symptom-directed PE. Results of physical examination will be presented in a listing and summarized by body system and by visit. Values out of the normal range judged by an Investigator as CS will be considered AEs.

# 12. INTERIM ANALYSES AND DATA SAFETY MONITORING

No interim analysis is planned for this study.

# 13. CHANGES TO PROTOCOL-SPECIFIED ANALYSES

There are no changes to protocol or to specified analyses for this study.

#### 14. GENERAL INFORMATION RELATED TO DATA PRESENTATIONS

All programs used to generate statistical analyses will be validated according to Algorithme Pharma's standard operating procedures.

Tables, Figures, and Listings (TFLs) will be displayed on letter size paper, 8 ½ inches by 11 inches, using the Courier New font.

In general, summary statistics for raw variables (i.e., variables measured at the study site or central laboratory) will be displayed as follows: minima and maxima will be displayed to the same number of decimal places as the raw data. Means, medians, and quartiles will be displayed to one additional decimal place and standard deviations will be displayed to two additional decimal places.

Percentages will be displayed to one decimal place. Percentages between 0 and 0.1 (exclusive) will be displayed as '<0.1'. P-values will be displayed to 3 decimal places. P-values that are less than 0.001 will be displayed as '<0.001'.

The numbers of decimal places for summary statistics of derived variables (i.e., variables that are not measured by the study site but are calculated for analysis based on other measured variables) will be determined on a case by case basis. In general, minima and maxima will be displayed to the commonly used unit of precision for the parameter. Means, medians, quartiles, and confidence limits will be displayed to one additional decimal place and standard deviations will be displayed to two additional decimal places.

The formats and layouts of TFLs are provided in subsequent sections. Actual formats and layouts may be altered slightly from those presented in the templates as necessary to accommodate actual data or statistics. Minor format changes will not require updates to the SAP.

# **PLANNED TABLES**

# **Demographic Data**

| Table 14.1.1 | Subject Disposition (All Subjects) |
|---|---|
| Table 14.1.2 | Demographic Characteristics by Analysis Population (Safety Population, Evaluable Population, PK Population) |
| Table 14.1.3 | Reasons for Subjects not Dosed (All Subjects) |
| Table 14.1.4 | Protocol Deviations (Safety Population) |
| Table 14.1.5 | Study Drug Exposure by Analysis Population (Safety Population, Evaluable Population, PK Population) |
| Table 14.1.6 | HAV Ribonucleic Acid (RNA) at Screening (Safety Population) |
| Table 14.1.7 | Prior Medications (Safety Population) |
| Table 14.1.8 | Concomitant Medications(Safety Population) |

# **PK Data**

| Table 14.2.1 | Percentage of Subjects Maintaining Anti-HAV Antibody Levels ≥10 mIU/mL up to Day 60 by Analysis Population (Safety Population and Evaluable Population) |
|---|---|
| Table 14.2.2.1 | Anti-HAV antibody Serum Baseline Uncorrected Concentrations by Analysis Population (Safety Population, Evaluable Population, PK Population) |
| Table 14.2.2.2 | Anti-HAV antibody Serum Baseline Corrected Concentrations by Analysis Population (Safety Population, Evaluable Population, PK Population) |
| Table 14.2.3.1 | Baseline Uncorrected PK parameters of Anti-HAV Antibody (PK Population) |
| Table 14.2.3.2 | Baseline Corrected PK Parameters of Anti-HAV Antibody (PK Population) |

# **Safety Data**

Tables in this section are based on the safety population unless otherwise stated.

| Table 14.3.1.1 | Overall Treatment-Emergent Adverse Events |
|---|---|
| Table 14.3.1.2.1 | Non-Treatment-Emergent Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.1.2.2 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.1.3 | Treatment-Emergent Adverse Events by Relationship to Study Drug |
| Table 14.3.1.4 | Suspected Adverse Drug Reactions by System Organ Class and Preferred Term |
| Table 14.3.1.5 | Treatment-Emergent Adverse Events by Severity |
| Table 14.3.1.6 | Treatment-Emergent Adverse Events by Seriousness |
| Table 14.3.1.7 | Injection Site Reactions by Location |
| Table 14.3.1.8 | Injection Site Reactions by Severity |
| Table 14.3.1.9 | Temporally-Associated Adverse Events |
| Table 14.3.1.10 | Adverse Event Leading to Discontinuation |
| Table 14.3.2 | Deaths and Other Serious Adverse Events |
| Table 14.3.3.1 | Hematology |
| Table 14.3.3.2 | Chemistry |
| Table 14.3.3.3 | Urinalysis |
| Table 14.3.3.4 | Shift from Baseline for Hematology |

| Table 14.3.3.5 | Shift from Baseline for Chemistry |
|----------------|------------------------------------|
| Table 14.3.3.6 | Shift from Baseline for Urinalysis |
| Table 14.3.4 | Vital signs |

## PLANNED FIGURES

| Section 14.2.6 | Mean PK Figures |
|---|---|
| Figure 14.2.6.1.1 | Mean Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Linear Scale |
| Figure 14.2.6.1.2 | Mean Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale |
| Figure 14.2.6.1.3 | Mean Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Linear Scale |
| Figure 14.2.6.1.4 | Mean Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale |
| Figure 14.2.6.2.1 | Median Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Linear Scale |
| Figure 14.2.6.2.2 | Median Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale |
| Figure 14.2.6.2.3 | Median Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Linear Scale |
| Figure 14.2.6.2.4 | Median Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale |
| Figure 14.2.6.3.1 | Individual Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Linear Scale |
| Figure 14.2.6.3.2 | Individual Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale |
| Figure 14.2.6.3.3 | Individual Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Linear Scale |
| Figure 14.2.6.3.4 | Individual Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale |

# PLANNED LISTINGS

| Listing 16.2.1 | Study Disposition (All Subjects) |
|----------------|-----------------------------------------|
| Listing 16.22 | Protocol Deviations (Safety Population) |

29

| Analysis Populations |
|---|
| Demographic Characteristics (Safety Population) |
| Medical History (Safety Population) |
| Contraceptive Methods (Safety Population) |
| Investigational Product Administration (Safety Population) |
| Adverse Events (Safety Population) |
| Chemistry (Safety Population) |
| Hematology (Safety Population) |
| Urinalysis (Safety Population) |
| Coagulation (Safety Population) |
| Virus Safety (Serology and NAT) Lab (Safety Population) |
| Urine Drug Screen (Safety Population) |
| Pregnancy Test (Safety Population) |
| Prior and Concomitant Medications (Safety Population) |
| Physical Examination (Safety Population) |
| Vital Signs (Safety Population) |
| Electrocardiogram Assessments (Safety Population) |
| Individual PK Data: Anti-HAV antibody |
| <u> </u> |
| Individual Serum Baseline Uncorrected Concentration Data of Anti-HAV antibody by<br>Timepoint Following a Single 0.2 mL/kg Intramuscular injection Administration of<br>GamaSTAN in HAV-seronegative healthy subjects (Safety Population) |
| Individual Serum Baseline Corrected Concentration Data of Anti-HAV antibody by |
| Timepoint Following a Single 0.2 mL/kg Intramuscular injection Administration of |
| GamaSTAN in HAV-seronegative healthy subjects (Safety Population) |
| Individual Serum Baseline Uncorrected PK parameters of Anti-HAV antibody Following a |
| Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV- |
| seronegative healthy subjects (PK Population) |
| obiologative floatilly adoption (i.i.t.) opalation/ |
| Individual Serum Baseline Corrected PK parameters of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV- |



# **APPENDIX A**

STUDY SCHEDULES

| Visits Procedures and Evaluation | Screening<br>Visit Days -28<br>to -2 | Day -1 | Day 1a | Day 2 | PK Sampling Visits b Days 3, 4, 5, 7, 10, 14, 21, 28, 60, 79, 115 | Final Visit (Day 150)b/<br>Early Discontinuation<br>Visit |
|---|---|---|---|---|---|---|
| Informed consent | X | | | | | |
| Admission to clinical research unit | | X | | | | |
| Inclusion/exclusion criteria | X | | | | | |
| Continued eligibility verification | | X | | | | |
| Medical history & demographics | X | | | | | |
| Height and weight | X | | | | | |
| ECG | X | X | | | | |
| Full physical exam c | X | | | | | X |
| Symptom-directed physical exam | | X | | X | X (Days 5, 28, and 60 visits only) | |
| Vital signs d | X | X | X | | X (Days 5, 28, and 60 visits only) | X |
| Clinical lab assessments e | X | X | | | X (Days 5, 28, and 60 visits only) | X |
| Coagulation tests (INR, aPTT) | X | | | | | |
| Immunoglobulin A (IgA) | X | | | | | |
| Pregnancy test f | X | X | | | | |
| Urine alcohol and drug panel testing g | X | X | | | | |
| Virus safety testing h | X | | | | | |
| Virus safety retain samples i | | | X | | | X |
| IP injection | | | X | | | |
| Injection site evaluation | | | X | X | | |

| Visits Procedures and Evaluation | Screening<br>Visit Days -28<br>to -2 | Day -1 | Day 1a | Day 2 | PK Sampling Visits Days 3, 4, 5, 7, 10, 14, 21, 28, 60, 79, 115 | Final Visit (Day 150)ь/<br>Early Discontinuation<br>Visit |
|---|---|---|---|---|---|---|
| PK sampling (anti-HAV antibody level) | | | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X |
| Discharge from clinical research unit | | | | X | | |

- Collection of virus safety retain samples on Day 1 will be performed prior to study treatment administration. Vital signs will be measured prior to study drug injection, approximately 60 minutes (±10 minutes) and 12 hours (±10 minutes) after study treatment administration. Injection site evaluation will be performed approximately 60 minutes after study treatment administration. PK blood sampling on Day 1: prior to study drug injection, 60 minutes (±10 minutes) post study drug injection and 12 hours post study drug injection (a window of ±1 hour is permitted)
- PK sampling visits will be conducted as close as possible to the exact time points. The PK sampling visits: Day 2 (window of ±1 hour); Days 3, 4 and 5 (visits have a window of ±4 hours); Days 7, 10, and 14 (all 3 visits have a window of ±1 day); Days 21 and 28 (both visits have a window of ±2 days); Days 60, 79 and 115 (all 3 visits have a window of ±4 days); Day 150 (a window of ±7 days)
- <sup>c</sup> Full physical examination (excluding breast and genitourinary examination)
- d Vital signs include systolic blood pressure, diastolic blood pressure, body temperature, heart rate, respiratory rate
- <sup>e</sup> Clinical laboratory assessments will include hematology, chemistry, and urinalysis. Hematology panel: hemoglobin, hematocrit, platelets, red blood cell count, and white blood cell count (absolute and % with differential). Chemistry panel: Sodium, potassium, creatinine, BUN, calcium, LDH, AST, ALT, GGT, ALP, glucose, total bilirubin, direct and indirect bilirubin. Urinalysis panel: Microscopic evaluation is done only with cause, pH, protein, glucose, and blood.
- Dipstick urine pregnancy test at screening visit and on Day -1 administration.
- g Urine alcohol and drug panel testing (drug panel includes marijuana, opiates, cocaine, amphetamines, methamphetamines and benzodiazepines)
- Virus safety testing: HAV RNA, HBV DNA, HCV RNA, HIV-1 RNA and B19V DNA by NAT methods as well as HAV antibody differential (IgM/IgG), hepatitis B core antibody differential (IgM/IgG), hepatitis C antibody, HIV-1/-2 + Group O antibody and B19V antibody differential (IgM/IgG) testing by serological methods.
- Virus safety retain samples: serum and/or plasma samples for HAV RNA, HBV DNA, HCV RNA, HIV-1 RNA and B19V DNA testing by NAT methods as well as HAV antibody differential (IgM/IgG), hepatitis B core antibody differential (IgM/IgG), hepatitis C antibody, HIV-1/-2 + Group O antibody and B19V antibody differential (IgM/IgG) testing by serological methods will be collected on Day 1 prior to IP injection and at final visit (Day 150)/early discontinuation visit. These samples will be tested only if the subject exhibits clinical signs and symptoms consistent with HAV, HBV, HCV, HIV or B19V infection while participating in the study. Virus safety retain samples will be retained until all analyses in support of the study are complete.

# **APPENDIX B**

## TABLE SHELLS

GENERAL PROGRAMMING NOTE: The displayed of decimals will follow Section 14 of the SAP for efficacy and safety outputs.



Hepatitis A Pre-exposure Prophylaxis


Table 14.1.1 Subject Disposition (All Subjects)

| | | Overall |
|---|---|---|
| Subjects Included [N] | Screened [1]<br>Re-Screened | XX<br>XX |
| Subjects not Dosed [N] | | xx |
| Subjects Dosed [N] | | xx |
| Subjects Completed the Study [n(%)] | YES<br>NO | xx (xx.x)<br>xx (xx.x) |
| <pre>If No, Reason(s) of Study Discontinuation [n(%)]</pre> | Reason 1<br>Reason 2<br>Reason 3<br>Etc. | xx (xx,x)<br>xx (xx,x)<br>xx (xx,x)<br>xx (xx,x) |
| Number of Subjects Included in Each Analysis Population $[n(\%)]$ | Safety Population<br>Evaluable Population<br>Pharmacokinetic Population | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

Note: The percentages are calculated using the number of subjects dosed as denominator.

[1] Screened subjects include re-screened subjects.

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas



GC1703 (GamaSTAN) Hepatitis A Pre-exposure Prophylaxis Page 1 of x Grifols

Table 14.1.2

Demographic Characteristics by Analysis Population
(Safety Population, Evaluable Population, PK Population)

| | | Safety Population (N=XX) | Evaluable<br>Population<br>(N=XX) | Pharmacokinetion<br>Population<br>(N=XX) |
|---|---|---|---|---|
| Age (years) | N | XX | XX | XX |
| rige (years) | Mean (SD) | xx (xx.x) | XX (XX.X) | XX (XX.X) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| Gender [n(%)] | MALE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | FEMALE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Childbearing Potential [n(%)] (Female Only) | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity [n(%)] | HISPANIC OR LATINO | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | NOT HISPANIC OR LATINO | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | UNKNOWN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race [n(%)] | WHITE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | AMERICAN INDIAN OR ALASKA NATIVE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | ASIAN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | BLACK OR AFRICAN AMERICAN | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Weight (kg) | N | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| Height (cm) | N | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| Body Mass Index (kg/m²) | N | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |


Notes: Fertility status percentage is based on the number of female subjects in the analysis population.

Subjects can contribute to more than one race category.




### Table 14.1.3 Reasons for Subjects not Dosed (All Subjects)

| | | Overall |
|---|---|---|
| Subjects not Dosed [N] | | xx |
| If No, Reason(s) of not Dose [n] | SCREEN FAILURE (INCLU<br>CRITERIA) | JSION/EXCLUSION xx |
| | OTHER | xx |

PROGRAMMING NOTE: 'OTHER' will be presented only if at least one subject that not dose have another reason for not dose than screen failure


## Table 14.1.4 Protocol Deviations (Safety Population)

| | Overall |
|-----------------------------------------------|------------|
| Characteristics | (N=XX) |
| Number of Protocol Deviations | xxxx |
| Subjects with at Least One Protocol Deviation | xxx (xx.x) |
| Type of Protocol Deviation [1][2] | |
| Deviation Category #1 | XX (XX.X) |
| Deviation Category #2 | XX (XX.X) |
| Deviation Category #3 | xx (xx.x) |
| Number of Major Protocol Deviations | xxxx |
| Subjects with at Least One Major Protocol | xxxx |
| Deviation | |
| Type of Major Protocol Deviation [1][2] | |
| Deviation Category #1 | xx (xx.x) |
| Deviation Category #2 | xx (xx.x) |
| Deviation Category #3 | xx (xx.x) |

#### PROGRAMMING NOTE: the Deviation Category will be repoted in the raw protocol deviation file and could be incluse (but not limited to) Inclusion / Exclusion criteria, ICF, etc.

- [1] The denominator is the number of subjects in the Safety Population.
- [2] Options are not mutually exclusive to each other. At each level of summary, each subject is only counted once.


Table 14.1.5

Study Drug Exposure by Analysis Population
(Safety Population, Evaluable Population, PK Population)

| | | | Safety Population<br>(N=XX) | Evaluable<br>Population<br>(N=XX) | Pharmacokinetic<br>Population<br>(N=XX) |
|---|---|---|---|---|---|
| Total Volume Prep | pared | N | xx | XX | XX |
| ( | | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX, XX | XX, XX | XX, XX |
| Total Vo<br>Administrated (mL) | lume | N | xx | XX | XX |
| , | | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX, XX | XX, XX | XX, XX |
| Treatment Compliance (%) | | N | XX | XX | XX |
| | | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX, XX | XX, XX | XX, XX |
| Duration of Treat<br>Administration (min) | ment | N | XX | XX | xx |
| | | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | XX, XX | XX, XX | XX, XX |
| Injection site | Right Upper Arm | n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Left Upper Arm | n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Right Upper Thigh | n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Left Upper Thigh | n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Treatment Compliance is defined as the total volume administered / total volume prepared x 100%




Table 14.1.6

HAV Ribonucleic Acid (RNA) at Screening (Safety Population)

| | | Overall (N=XX) |
|----------|------|----------------|
| Positive | n(%) | xx (xx.x) |
| Negative | n(%) | xx (xx.x) |

PROGRAMMING NOTE: if the LBTEST=HCV Viral Load had a result showing 'NOT DETECTED', it will be considered as NEGATIVE; Otherwise, if the virus present a detected result, it will be considered as POSITIVE.




## Table 14.1.7 Prior Medications (Safety Population)

| ATC Level 2 / | |
|--------------------------|-----------|
| ATC Level 4 | Overall |
| | (N=XX) |
| Any Medication [n(%)] | xx (xx.x) |
| Classification #1 [n(%)] | |
| Medication #1* [n(%)] | xx (xx.x) |
| Medication #2 [n(%)] | xx (xx.x) |
| Medication #3 [n(%)] | xx (xx.x) |
| | xx (xx.x) |
| Classification #2 [n(%)] | |
| Medication #1 [n(%)] | xx (xx.x) |
| Medication #2 [n(%)] | xx (xx.x) |
| Medication #3 [n(%)] | xx (xx.x) |
| Etc. | xx (xx.x) |
| Etc. | |

Note(s): ATC= Anatomical Therapeutic Chemical.

Medication classifications are coded to ATC Levels 2 and 4 using WHO-DDE dictionary version March 1, 2017  $^{\star}$  The higher ATC level term is used if ATC Level 2 or 4 are missing.

The figure are level of the bound of the figure and the figure are the figure and the figure are the figure and the figure are the figure and the figure are

All medications stopped prior to the start of IP injection are included.

Each subject is only counted once at each level of summation.




# Table 14.1.8 Concomitant Medications (Safety Population)

| ATC Level 2 / | |
|--------------------------|-----------|
| ATC Level 4 | Overall |
| | (N=XX) |
| Any Medication [n(%)] | xx (xx.x) |
| Classification #1 [n(%)] | |
| Medication #1* [n(%)] | xx (xx.x) |
| Medication #2 [n(%)] | xx (xx.x) |
| Medication #3 [n(%)] | xx (xx.x) |
| | xx (xx.x) |
| Classification #2 [n(%)] | |
| Medication #1 [n(%)] | xx (xx.x) |
| Medication #2 [n(%)] | xx (xx.x) |
| Medication #3 [n(%)] | xx (xx.x) |
| Etc. | xx (xx.x) |
| Etc. | |

Note(s): ATC= Anatomical Therapeutic Chemical.

Medication classifications are coded to ATC Levels 2 and 4 using WHO-DDE dictionary version March 1, 2017

 $^{\star}$  The higher ATC level term is used if ATC Level 2 or 4 are missing.

All medications started on or after the start of IP injection, or taken prior to and continued after the start of IP injection are included.

Each subject is only counted once at each level of summation.

Table 14.2.1 Percentage of Subjects Maintaining Anti-HAV Antibody Levels  $\geq 10$  mIU/mL up to Day 60 by Analysis Population (Safety Population and Evaluable Population)

| | | Safety Population<br>(N=XX) | Evaluable<br>Population<br>(N=XX) |
|---|---|---|---|
| Subjects Maintaining Anti-HAV Antibody Levels $\geqslant 10$ mIU/mL up to Day 60 | n (%) | xx (xx.x) | xx (xx.x) |

Hepatitis A Pre-exposure Prophylaxis

Table 14.3.1.1 Overall Treatment-Emergent Adverse Events (Safety Population)

| | Statistic | Overall<br>(N=XX) |
|---|---|---|
| Subjects with Any Treatment-Emergent Adverse Events (TEAEs) | N (%) | xx (xx.x) |
| Total Number of TEAEs | N | xxx |
| Subjects with Suspected Adverse Drug Reactions (ADRs)[1] | N (%) | xx (xx.x) |
| Total Number of Suspected ADRs | N | xxx |
| Subjects with Adverse Reactions (ARs) [2] | N (%) | xx (xx.x) |
| Total Number of ARs | N | XXX |
| Subjects with Serious Adverse Events (SAEs) | N (%) | xx (xx.x) |
| Total Number of SAEs | N | xxx |
| Subjects with TEAEs Leading to Discontinuation from Study | N (%) | xx (xx.x) |
| Total Number of TEAEs Leading to Discontinuation | N | xxx |
| Subjects with TEAEs with Outcome of Death | N (%) | xx (xx.x) |
| Total Number of Deaths | N | xxx |
| Subjects with Injection Site Reactions | N (%) | xx (xx.x) |
| Total Injection Site Reactions | N | xxx |
| Subjects with TEAEs during/within 24 Hours post IP Injection | N (%) | xx (xx.x) |
| Total Number of TEAEs during/within 24 Hours post IP Injection | N | xxx |
| Subjects with TEAEs during/within 72 Hours post IP Injection | N (%) | xx (xx.x) |
| Total Number of TEAEs during/within 72 Hours post IP Injection | N | XXX |

<sup>[1]</sup> A suspected adverse drug reaction is an adverse event with investigator's causality assessment of 'definitely related' or 'possibly related'.

<sup>[2]</sup> An adverse reaction is a suspected adverse drug reaction with a causal relationship of "definitely related".

Data Source: XXXX Program Source: XXXXX.sas

Date: VERSION - YYYY-MM-DD Data Source: XXXX

 ${\tt Table~14.3.1.2.2}$   ${\tt Treatment-Emergent~Adverse~Events~by~System~Organ~Class~and~Preferred~Term} \end{\ensuremath} \begin{tabular}{ll} (Safety~Population) \end{\ensuremath}$ 

| | | Overall | |
|----------------------|-----------|-----------|-----------|
| System Organ Class / | Statistic | Subjects | Events |
| Preferred Term | | (N=XX) | (N=XX) |
| Any TEAEs | N (%) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | | | |
| Preferred Term 1 | N (%) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | N (%) | xx (xx.x) | xx (xx.x) |
| System Organ Class 2 | | | |
| Preferred Term 1 | N (%) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | N (%) | xx (xx.x) | xx (xx.x) |

Notes: Adverse Events are coded using MedDRA, version 20.1.

At each level of summation, each subject is counted only once.

'N' for events in the column headers is the total number of TEAEs and is used as the denominator for all % in that column.

#### Similar Tables

Table 14.3.1.2.1 Non-Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

Table 14.3.1.4 Suspected Adverse Drug Reactions by System Organ Class and Preferred Term
PROGRAMMING NOTE: Note:] A suspected adverse drug reaction is an adverse event with investigator's causality assessment of 'definitely related' or 'possibly related'.

Table 14.3.1.3

Treatment-Emergent Adverse Events by Relationship to Study Drug (Safety Population)

| · | · | · | Overa | 111 |
|---|---|---|---|---|
| System Organ Class / | | Statistic | Subjects | Events |
| Preferred Term | | | (N=XX) | (N=XX) |
| Any TEAEs | Unrelated/Not Related | N (%) | xx (xx.x) | xx (xx.x) |
| | Possibly Related | N (%) | xx (xx.x) | xx (xx.x) |
| | Definitely Related | N (%) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | Unrelated/Not Related | N (%) | xx (xx.x) | xx (xx.x) |
| | Possibly Related | N (%) | xx (xx.x) | xx (xx.x) |
| | Definitely Related | N (%) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | Unrelated/Not Related | N (%) | xx (xx.x) | xx (xx.x) |
| | Possibly Related | N (%) | xx (xx.x) | xx (xx.x) |
| | Definitely Related | N (%) | xx (xx.x) | xx (xx.x) |

Notes: Adverse Events are coded using MedDRA, version 20.1.

At each level of summation by subject (Overall, System Organ Class, and Preferred Term), each subject is only counted once under the greatest causality.

Table 14.3.1.5

Treatment-Emergent Adverse Events by Severity
(Safety Population)

| | | | Overall | |
|----------------------|----------|-----------|-----------|-----------|
| System Organ Class / | | Statistic | Subjects | Events |
| Preferred Term | | | (N=XX) | (N=XX) |
| Any TEAEs | Mild | N (%) | xx (xx.x) | xx (xx.x) |
| | Moderate | N (%) | xx (xx.x) | xx (xx.x) |
| | Severe | N (%) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | Mild | N (%) | xx (xx.x) | xx (xx.x) |
| | Moderate | N (%) | xx (xx.x) | xx (xx.x) |
| | Severe | N (%) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | Mild | N (%) | xx (xx.x) | xx (xx.x) |
| | Moderate | N (%) | xx (xx.x) | xx (xx.x) |
| | Severe | N (%) | xx (xx.x) | xx (xx.x) |

Notes: Adverse Events are coded using MedDRA, version 20.1.

At each level of summation by subject (Overall, System Organ Class, and Preferred Term), each subject is only counted once under the greatest severity.

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

Similar Table:

Table 14.3.1.8 Injection Site Reactions by Severity

Table 14.3.1.6
Treatment-Emergent Adverse Events by Seriousness (Safety Population)

| | | | Overall | |
|----------------------|-------------|-----------|-----------|-----------|
| System Organ Class / | | Statistic | Subjects | Events |
| Preferred Term | | | (N=XX) | (N=XX) |
| Any TEAEs | Serious | N (%) | xx (xx.x) | xx (xx.x) |
| | Not Serious | N (%) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | Serious | N (%) | xx (xx.x) | xx (xx.x) |
| | Not Serious | N (%) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | Serious | N (%) | xx (xx.x) | xx (xx.x) |
| | Not Serious | N (%) | xx (xx.x) | xx (xx.x) |

Notes: Adverse Events are coded using MedDRA, version 20.1.

At each level of summation by subject (Overall, System Organ Class, and Preferred Term), each subject is only counted once, and being serious has higher priority than not serious

Table 14.3.1.7
Injection Site Reactions by Location (Safety Population)

| | | | Overa | 111 |
|----------------------|-------------------|-----------|-----------|-----------|
| System Organ Class / | | Statistic | Subjects | Events |
| Preferred Term | | | (N=XX) | (N=XX) |
| Any TEAEs | Right Upper Arm | N (%) | xx (xx.x) | xx (xx.x) |
| | Left Upper Arm | N (%) | xx (xx.x) | xx (xx.x) |
| | Right Upper Thigh | N (%) | xx (xx.x) | xx (xx.x) |
| | Left Upper Thigh | N (%) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | Right Upper Arm | N (%) | xx (xx.x) | xx (xx.x) |
| | Left Upper Arm | N (%) | xx (xx.x) | xx (xx.x) |
| | Right Upper Thigh | N (%) | xx (xx.x) | xx (xx.x) |
| | Left Upper Thigh | N (%) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | Right Upper Arm | N (%) | xx (xx.x) | xx (xx.x) |
| | Left Upper Arm | N (%) | xx (xx.x) | xx (xx.x) |
| | Right Upper Thigh | N (%) | xx (xx.x) | xx (xx.x) |
| | Left Upper Thigh | N (%) | xx (xx.x) | xx (xx.x) |

Notes: Adverse Events are coded using MedDRA, version 20.1.

At each level of summation by subject (Overall, System Organ Class, and Preferred Term), each subject is only counted once under each location.

Table 14.3.1.9
Temporally-Associated Adverse Events
(Safety Population)

| | | | | Overa | 11 |
|---|---|---|---|---|---|
| System Organ Class / | | | Statistic | Subjects | Events |
| Preferred Term | | | | (N=XX) | (N=XX) |
| Any TEAEs | During/Within 24 hours Injection | Post | N (%) | xx (xx.x) | xx (xx.x) |
| | During/Within 72 hours<br>Injection | Post | N (%) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | During/Within 24 ho<br>Injection | urs Post | N (%) | xx (xx.x) | xx (xx.x) |
| | During/Within 72 ho<br>Injection | urs Post | N (%) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | During/Within 24 ho<br>Injection | urs Post | N (%) | xx (xx.x) | xx (xx.x) |
| | During/Within 72 ho<br>Injection | urs Post | N (%) | xx (xx.x) | xx (xx.x) |

Notes: Adverse Events are coded using MedDRA, version 20.1.

At each level of summation by subject (Overall, System Organ Class, and Preferred Term), each subject is only counted once for each duration.

A temporally-associated AEs is defined as AEs happening during IP injection or within 24 hours following the end of IP Injection and within 72 hours following the end of IP injection

Similar Table:

Table 14.3.1.10 Adverse Events Leading to Discontinuation


### Table 14.3.2 Deaths and Other Serious Adverse Events (Safety Population)

| | | | | | Resolution | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | SOC/ | | | Date | | | | |
| | Injection | | | | Time | | | | |
| | site | Prefe | | | (Time since | | | | |
| | reaction?/ | rred | Onset I | ate | Start of | S: | | A: Action Taken with | |
| | Injection | Term/ | Time | | Study | Severity | | Study Treatment | If |
| | Site | | (Time si | nce | Treatment | R: | O: Outcome | ANDT: Additional | any, |
| | Reaction | Descr | Start | of | [1]) | Relations | S: Serious AE | Non-Drug Treatment | Reason |
| | Location | iptio | Study | | (AE | hip to IP | D: AE leading | TRT: Specify | for |
| Subject | / | n of | Treatmen | t[1 | Duration | F: | to Study | treatment | Seriou |
| ID | AE # | AE | ]) | | [2])) | Frequency | Discontinuation | C: Concomitant Given | sness |

PROGRAMMING NOTE: Subject with SAE or ar least one Reason for Seriousness or dead will be included in this listing

Notes: Adverse Events are coded using MedDRA, version 20.1.

- [1] Time since start of study treatment is presented in days if >24 hours or in hh:mm if <=24 hours.
- [2] AE duration is presented in days if >24 hours or in hh:mm if <=24 hours.

Table 14.3.3.1 Hematology (Safety Population)

| | | | | | verall<br>N=XX) |
|---|---|---|---|---|---|
| | | | | Actual Value | Change from Baseline |
| Parameter (unit) | Visit | | | notaal varat | onango IIom DasoIImo |
| Lab Test 1 | | | | | |
| | XXX | Value | N | xx | |
| | | | Mean (SD) | xx (xx.x) | |
| | | | Median | XX.X | |
| | | | Min, Max | XX, XX | |
| | | | IQR | xx; xx | |
| | XXX | Value | N | xx | |
| | | | Mean (SD) | xx (xx.x) | |
| | | | Median | XX.X | |
| | | | Min, Max | XX, XX | |
| | | | IQR | xx; xx | |
| | XXX | Value | N | XX | xx |
| | | | Mean (SD) | xx (xx.x) | xx (xx.x) |
| | | | Median | XX.X | XX.X |
| | | | Min, Max | XX, XX | XX, XX |
| | | | IQR | xx; xx | xx; xx |
| | Etc | | | | |
| Etc | | | | | |

Similar Table:

Table 14.3.3.2 Chemistry Table 14.3.3.3 Urinalysis

Table 14.3.3.4
Shift from Baseline for Hematology (Safety Population)

| | | | | Baseline Result | | |
|---|---|---|---|---|---|---|
| | Post-Baseline | | Low | Normal | High | Total |
| Parameter (unit) | Visit | Result | n(%) | n(%) | n(%) | n(%) |
| XXXX | XXXX | Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): Only patients with a baseline result and post-baseline visit result are included.

For each parameter, percentages are based on total number of subjects with available results at both the baseline and the corresponding visit.

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

#### Similar Table:

Table 14.3.3.5 Shift from Baseline for Chemistry Table 14.3.3.6 Shift from Baseline for Urinalysis

Table 14.3.4 Vital Signs (Safety Population)

| | | | | | Over | |
|---|---|---|---|---|---|---|
| Parameter (unit) | Visit | Timepoint | | Actual Value | Change from<br>Baseline | |
| Systolic Blood<br>Pressure (mmHg) | XXX | | Value | N | XX | |
| Toodaro (mming) | | | | Mean (SD) | xx (xx.x) | |
| | | | | Median | XX.X | |
| | | | | Min, Max | XX, XX | |
| | XXX | | Value | N | XX | |
| | | | | Mean (SD) | xx (xx.x) | |
| | | | | Median | XX.X | |
| | | | | Min, Max | XX, XX | |
| | XXX | Pre-Dose | Value | N | XX | |
| | | | | Mean (SD) | xx (xx.x) | |
| | | | | Median | XX.X | |
| | | | | Min, Max | XX, XX | |
| | | 60 Minutes Post-Dose | Value | N | XX | XX |
| | | | | Mean (SD) | xx (xx.x) | xx (xx.x) |
| | | | | Median | XX.X | XX.X |
| | | | | Min, Max | XX, XX | XX, XX |
| | Etc. | | | | | |
| Etc. | | | | | | |
| PROGRAMMING NOTE: A | All visit | s outlined in Appendix A | A will be included. | | | |

#### **APPENDIX C**

LISTING SHELLS


Listing 16.2.1 Study Disposition (All Subjects)

| | Re-Screened | | Date of | | | | |
|---|---|---|---|---|---|---|---|
| | Subject? | / | Completion or | | | | |
| | Previous | | Discontinuatio | | | | |
| Subject ID | Subject ID | | n (Study Day) | Subject Status | Specify | AE # | Date of Death |

Note: Study Day is relative to the start of study treatment.

Page 1 of x GC1703 (GamaSTAN) Grifols

Hepatitis A Pre-exposure Prophylaxis

Listing 16.2.2 Protocol Deviations (Safety Population)

| | Deviation | | Deviation | Seve | | St | art Da | te (Study |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Category | Description | Criteria | ity | Action Taken | Da | 7) | |

Note: Study Day is relative to the start of study treatment.

Data Source: XXXX Program Source: XXXXX.sas Date: VERSION - YYYY-MM-DD

Listing 16.2.3 Analysis Populations

| | | | Reason |
|---|---|---|---|
| | | | of |
| | | | Exclusi |
| | | | on of |
| | | | the |
| | | | Evaluab |
| | | Reason of Exclusion | le PK |
| | | of the Safety | Populat Populatio Reason of Exclusion of |
| Subject ID | Safety Population | Population Evaluable Population | ion n the PK population |

Listing 16.2.4.1
Demographic Characteristics
(Safety Population)

| | | | Race/ | |
|---|---|---|---|---|
| Age | | | Other | |
| Subject ID (years) | Gender | Ethnicity | Race | Weight (kg) Height (cm) BMI (kg/m²) |

Listing 16.2.4.2 Medical History (Safety Population)

| | | | | C<br>urrently<br>taking<br>medicatio | | | | |
|---|---|---|---|---|---|---|---|---|
| | | SOC | Start<br>Date | n for<br>this | | | | |
| Subject<br>ID | MH # | Preferred Term Description of MH | (Study<br>Day) | condition ? | End Date | (Study Day) | MD Safety | Review [1] |

[1] NCS: Not Clinically Significant / CS: Clinically Significant

Note: Medical History is classified using MedDRA, version 20.1. Study Day is relative to the start of study treatment.


Listing 16.2.4.3 Contraceptive Methods (Safety Population)

Subject ID Category Contraceptive Method

PROGRAMMING NOTE: The category will correspond to Childbearing Potential, Birth Control Method and Non-Childbearing Birth Control Method

Date: VERSION - Data Source: XXXXX Program Source: XXXXX.sas

YYYY-MM-DD

### Listing 16.2.5 Investigational Product Administration (Safety Population)

| Subject | Start Date/Time | End Date/Time | | Desc | Double of | Thiogtion | ume<br>Adm<br>ini | Volumn<br>e<br>Admini<br>stered<br>per<br>Inject<br>ion | Nee<br>dle | Total volume Prepar ed (mL)/T otal Volume Admini | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjec | (Study | (Study | | Dose | Route of | Injection | ste | Site | Siz | stered | |
| t ID Visit | Day) | Day) | Treatment | Administered | Administration | Site | red | (mL) | e | (mL) | Comment |

Note: Percentage of Volume Administered is defined as follow: (Volume Administered (mL) / Volume Prepared (mL) \*100 Study Day is relative to the start of study treatment.


Listing 16.2.7 Adverse Events (Safety Population)

| | | | | | | | A: Action Taken | |
|---|---|---|---|---|---|---|---|---|
| | | | | Resolution | | | A: ACCION TAKEN | |
| | Injection | | | Date | | | with Study | |
| | site | | Onset Date | Time | | | Treatment | |
| | reaction?/ | | Time | (Time since | | | ANDT: | |
| | Injection | | (Time | Start of | | | Additional Non- | |
| | Site | SOC/ | since | Study | | O: Outcome | Drug Treatment | If any, |
| | Reaction | Preferred | Start of | Treatment | S: Severity | S: Serious AE | TRT: Specify | Reason |
| | Location | Term/ | Study | [1]) | R: Relationship | D: AE leading to | treatment | for |
| Subject | / | Description | Treatment | (AE Duration | to IP | Study | C: Concomitant | Serious |
| ID | AE # | of AE | [1]) | [2]) | F: Frequency | Discontinuation | Given | ness |

Note: Adverse Events as coded using MedDRA, version 20.1.

- [1] Time since start of study treatment is presented in days if >24 hours or in hh:mm if <=24 hours.
- [2] AE duration is presented in days if >24 hours or in hh:mm if <=24 hours.

Date: VERSION - YYYY-MM-DD Data Source: XXXX

Program XXXXX.sas Source:

Listing 16.2.8.1 Chemistry (Safety Population)

| | | | Parame | | | | |
|---|---|---|---|---|---|---|---|
| | | Collection | ter | Reference | | | |
| Subject ID | Visit | | (Unit) | Range | Value | Change From Baseline | Flag |

Date: VERSION - YYYY-MM-DD Data Source: XXXX

L16.2.8.2 Hematology
L16.2.8.3 Urinallysis
L16.2.8.4 Coagulation
L16.2.8.5 Virus Safety (Serology and NAT) Lab
L16.2.8.6 Urine Drug Screen
L16.2.8.7 Pregnancy Test


## Listing 16.2.8.8 Prior and Concomitant Medications (Safety Population)

| | CM#/ | | | | | | | | Start | End |
|---|---|---|---|---|---|---|---|---|---|---|
| | Prior or | Related | to ATC Level 2 / | | | | | | Date/Time | Date/Time |
| Subject | Concomit | AE#/ | ATC Level 4 / | | | | | | (Study | (Study |
| ID | nat? | MH# | Medication Name | Indication | Dose (unit) | Frequency | Formulation | Route | Day) | Day) |

Note: Medication classifications are coded to ATC Levels 2 and 4 using the WHO-DDE dictionary, Version March 1, 2017. The higher ATC level term is used if ATC Level 2 or 4 are missing.

Study Day is relative to the start of study treatment.

Listing 16.2.8.9
Physical Examination
(Safety Population)

Subject ID Visit Date/Time Assessment Result (Abnormal Findings) [1]

[1] NCS: Not Clinically Significant / CS: Clinically Significant

Listing 16.2.8.10
Vital Signs
(Safety Population)

| | | | | Assessment | | Change Fro | m Safety |
|---|---|---|---|---|---|---|---|
| Subject ID | Visit | Position | Date/Time | (Unit) | Range Value | Baseline | Review [1] |

[1] NCS: Not Clinically Significant / CS: Clinically Significant
GC1703 (GamaSTAN)

Hepatitis A Pre-exposure Prophylaxis

Grifols

Listing 16.2.8.11
Electrocardiogram Assessments
(Safety Population)

| Subject ID | Visit | Date/Time | Position | Parameter (Unit) | Result[1] |
|---|---|---|---|---|---|
| | | YYYY-MM- | | | |
| XXXXX | XXXXXX | DD/HH:MM | XXXXXX | ECG Parameter 1 | XX. X |
| | | | XXXXXX | ECG Parameter 2 | XX.X |
| | | | XXXXXX | Etc. | XX.X |
| | | | | Interpretation | XX.X |
| | | YYYY-MM- | | | |
| | | DD/HH:MM | XXXXXX | xxxxxx | XX.X |
| | | YYYY-MM- | | | |
| | | DD/HH:MM | XXXXXX | XXXXXX | XX.X |
| | | YYYY-MM- | | | |
| XXXXX | XXXXXX | DD/HH:MM | XXXXXX | XXXXXX | XX.X |
| ******** | ********** | 22, 1111 1111 | ********** | ********** | ***** |
| | | YYYY-MM- | | | |
| XXXXX | XXXXXX | DD/HH:MM | XXXXXX | Xxxxxx | XX.X |

[1] NCS: Not Clinically Significant / CS: Clinically Significant

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

## **APPENDIX D**

# SHELLS (FROM WINNONLIN)

Table 14.2.2.1 Anti-HAV antibody Serum Baseline Uncorrected Concentrations by Analysis Population (Safety Population, Evaluable Population, PK Population)

| Population | Parameter | Pre Injection | 1Hour | 12 Hours | 24 Hours | 48 Hours | <br>2736 Hours | 3576 Hours |
|---|---|---|---|---|---|---|---|---|
| Safety Population | N | l | | L | L | L | | |
| | Mean | | | | | | | |
| | SD | | | | | | | |
| | Min | | | | | | | |
| | Median | | | | | | | |
| | Max | | | | | | | |
| | CV% | | | | | | | |
| | CI 90% Lower | | | | | | | |
| | CI 90% Upper | | | | | | | |
| | Geometric Mean | | | | | | | |
| Evaluable Population | N | | | | | | | |
| | Mean | | | | | | | |
| | SD | | | | | | | |
| | Min | | | | | | | |
| | Median | | | | | | | |
| | Max | | | | | | | |
| | CV% | | | | | | | |
| | CI 90% Lower | | | | | | | |
| | CI 90% Upper | | | | | | | |
| | Geometric Mean | | | | | | | |

| PK Population | N N |
|---------------|----------------|
| | Mean |
| | SD |
| | Min |
| | Median |
| | Max |
| | CV% |
| | CI 90% Lower |
| | CI 90% Upper |
| | Geometric Mean |

Similar Table(s): Table 14.2.2.2 Anti-HAV antibody Serum Baseline Corrected Concentrations by Analysis Population (Safety Population, Evaluable Population, PK Population)

Table 14.2.3.1 Baseline Uncorrected PK parameters of Anti-HAV Antibody (PK Population)

| Parameter | AUC <sub>0-∞</sub> | AUC <sub>0-T</sub> | C <sub>max</sub> | $T_{max}$ | T <sub>half</sub> | CI <sub>тот</sub> /F | V <sub>D</sub> /F | λz |
|---|---|---|---|---|---|---|---|---|
| N | | | | | | | | |
| Mean | | | | | | | | |
| SD | | | | | | | | |
| Min | | | | | | | | |
| Median | | | | | | | | |
| Max | | | | | | | | |
| CV% | | | | | | | | |
| Geometric Mean | | | | | | | | |
| CV% Geometric Mean | | | | | | | | |
| CI 90% Lower | | | | | | | | |
| CI 90% Upper | | | | | | | | |
| CI 90% Lower GEO Mean | | | | | | | | |
| CI 90% Upper GEO Mean | | | | | | | | |

Similar Table(s): Table 14.2.3.2 Baseline Corrected PK parameters of Anti-HAV Antibody (PK Population)

Listing 16.2.6.1 Individual Serum Baseline Uncorrected Concentration Data of Anti-HAV antibody by Timepoint Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (Safety Population)

| Subject | Scheduled Timepoint Date | Scheduled Timepoint Date Time Nominal Time Actual Elapse (units) (units) | - |
|---|---|---|---|

## Similar Listing(s)

Listing 16.2.6.2 Individual Serum Baseline Corrected Concentration Data of Anti-HAV antibody by Timepoint Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (Safety Population)

Listing 16.2.6.3 Individual Serum Baseline Uncorrected PK parameters of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population)

| Subject | AUC <sub>0-∞</sub><br>(units) | AUC <sub>0-T</sub><br>(units) | C <sub>max</sub><br>(units) | T <sub>max</sub><br>(units) | T <sub>half</sub><br>(units) | CI <sub>TOT</sub> /F<br>(units) | V <sub>D</sub> /F<br>(units) | Λz<br>(units) |
|---|---|---|---|---|---|---|---|---|

Listing 16.2.6.3 Individual Serum Baseline Uncorrected PK parameters of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) (Cont'd)

| Subject | Number of Point | R² | T <sub>LIN</sub><br>(Unit) | T <sub>LQC</sub><br>(unit) | AUC <sub>%Extrap</sub> (Unit) |
|---|---|---|---|---|---|

Similar Listing(s):

Listing 16.2.6.4 Individual Serum Baseline Corrected PK parameters of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population)

Section 14.2.6 Mean PK Figures

Figure 14.2.6.1.1 Mean Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) - Linear Scale



## Similar Figure(s):

- Figure 14.2.6.1.3 Mean Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) Linear Scale
- Figure 14.2.6.2.1 Median Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) Linear Scale
- Figure 14.2.6.2.3 Median Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) Linear Scale

Figure 14.2.6.1.2 Mean Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale



Note: The figures do not reflect the actual data of the study.

## Similar Figure(s):

Figure 14.2.6.1.4 Mean Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale

Figure 14.2.6.2.2 Median Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale

Figure 14.2.6.2.4 Median Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale

Figure 14.2.6.3.1 Individual Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Linear Scale



Similar Figure(s):

Figure 14.2.6.3.3 Individual Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Linear Scale

Figure 14.2.6.3.2 Individual Serum Baseline Uncorrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale



Similar Figure(s):

Figure 14.2.6.3.4 Individual Serum Baseline Corrected Concentration-Time Profile of Anti-HAV antibody Following a Single 0.2 mL/kg Intramuscular injection Administration of GamaSTAN in HAV-seronegative healthy subjects (PK Population) – Semi-Log Scale



Study Number: GC1703 26 Nov 2018

Study Number: GC1703 GamaSTAN®: Clinical Study Report

# 16.1.9.2 Statistical Output

Not applicable.